CLINICAL TRIAL: NCT06558799
Title: LUNAR-4: Pilot, Single Arm, Open-Label, Multinational Study of Tumor Treating Fields (TTFields, 150 kHz) Concomitant With Pembrolizumab for the Treatment of Metastatic Non-Small Cell Lung Cancer (NSCLC) Previously Treated With a PD-1/PD-L1 Inhibitor and Platinum-Based Chemotherapy
Brief Title: LUNAR-4: Effect of Tumor Treating Fields (TTFields) (150 kHz) Concurrent With Pembrolizumab for Treatment of Metastatic Non-small Cell Lung Cancer (NSCLC)
Acronym: LUNAR-4
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NovoCure GmbH (Industry)
Responsible Party: Sponsor
Organization: NovoCure Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF-50
Record Dates: First submitted 2024-07-31; First posted 2024-08-19 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; Metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- NovoTTF-200T + Pembrolizumab (Experimental)
  Interventions: Device: NovoTTF-200T; Drug: Pembrolizumab

INTERVENTIONS:
Device: NovoTTF-200T — The NovoTTF-200T is a portable, battery operated system intended for continuous home use, which delivers TTFields at a frequency of 150kHz to the subject by means of insulated transducer arrays. TTFields exert electric forces intended to disrupt cancer cell division and induce immunogenic cell death.
Drug: Pembrolizumab — Pembrolizumab is an immune checkpoint inhibitor that helps the immune system recognize and attack cancer cells.

SUMMARY:
The purpose of the study is to test the effectiveness and safety of TTFields therapy, delivered using the NovoTTF-200T device, concomitant with pembrolizumab in subjects with metastatic NSCLC previously treated with a PD-1/PD-L1 inhibitor and platinum-based chemotherapy.

ELIGIBILITY:
INCLUSION CRITERIA:

* ≥18 years of age
* Histologically or cytologically confirmed diagnosis of NSCLC.
* Documented positive tumor PD-L1 expression (TPS≥1%).
* Eastern Cooperative Oncology Group (ECOG) Score of 0-1.
* Diagnosis of radiological progression while on or after first platinum-based systemic therapy administered for advanced or metastatic disease.
* Subjects must have received one line of PD-1/PD-L1 inhibitor therapy for advanced or metastatic NSCLC. PD-1/PD-L1 inhibitor may have been given alone or in combination with other therapy.
* Subjects who received PD-1/PD-L1 inhibitor for advanced disease, must have had a best response on PD-1/PD-L1 inhibitor of stable disease (SD), partial response (PR) or complete response (CR).
* Subjects must have experienced disease progression more than 84 days following Cycle 1 Day 1 (C1D1) of their most recent PD-1/PD-L1 inhibitor therapy.

EXCLUSION CRITERIA - All individuals meeting any of the following exclusion criteria will be excluded from study participation:

* Mixed small cell and NSCLC histology.
* Subject must not have leptomeningeal disease or spinal cord compression.
* Subject must not have untreated, symptomatic brain metastases, or residual neurological dysfunction.
* Subjects must not have received more than one line of PD-1/PD-L1 inhibitor for advanced disease.
* Subjects with a known sensitizing mutation for which the Food and Drug Administration (FDA)-approved targeted therapy for NSCLC exists (e.g., EGFR, ALK, ROS1) are excluded unless previously received at least one of the approved therapy(ies).
* Subjects with more than 2 lines of therapy in the advanced setting.
* Pregnant or breastfeeding.
* Implantable electronic medical devices (e.g. pacemaker, defibrillator) in the upper torso.
* Known allergies to medical adhesives or hydrogel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 16
  To compare OS in subjects treated with TTFields concomitant with pembrolizumab compared to OS of subjects who were treated with docetaxel alone in the LUNAR/ EF-24 study (superiority analysis)

CONTACTS AND LOCATIONS:
Locations (24):
- Universitätsklinik f. Innere Medizin III, Salzburg, Austria
- Czechia (3):
  - Vitkovicka Nemocnice, Ostrava
  - General University Hospital in Prague, Clinic of Oncology, Prague
  - FN Motol, Prague
- France (7):
  - APHP - Hôpital Ambroise-Paré, Boulogne-Billancourt
  - Centre hospitalier intercommunal de Créteil Service de Pneumologie, Créteil
  - Centre Léon Berard Service D'oncologie Médicale, Lyon
  - Hôpital Européen Marseille, Marseille
  - Montpellier University Hospital, Montpellier
  - Hôpital Privé du Confluent Service D'oncologie Médicale, Nantes
  - Centre Hospitalier Intercommunal de Cornouaille Service D'oncologie Médicale, Quimper
- Italy (4):
  - Humanitas Gavazzeni Bergamo-U.O.Farmacia-Edificio D Piano -1, Bergamo
  - Istituto Europeo di Oncologia, Milan
  - AO SM Misericordia di Perugia, Perugia
  - AOUS Policlinico Le Scotte U.O.C. Immunoterapia Oncologica, Siena
- Rijnstate Ziekenhuis, Arnhem, Netherlands
- Poland (2):
  - Pratia MCM Kraków, Krakow
  - MS Pneumed Janusz Milanowski, Katarzyna Szmygin-Milanowska Spó?ka Jawna, Lublin
- Spain (6):
  - Hospital Universitario del Vinalopó, Elche
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Clínica Universidad de Navarra, Madrid, Madrid
  - Hospital Regional Universitario de Malaga (Hospital Civil), Málaga
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocio, Seville